CLINICAL TRIAL: NCT05725421
Title: Oncologic, Functional and Surgical Outcomes for Patients Undergoing Radical Nephrectomy for Low-Risk Renal Cell Carcinoma and Recipients of Reconstructed Renal Allografts Following Ex-Vivo Partial Nephrectomy
Brief Title: Transplantation of Reconstructed Renal Allografts Following Ex-Vivo Partial Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE13822
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Radical Nephrectomy; Renal Allograft; Ex-Vivo Partial Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cT1a Radical Nephrectomy + Donor Kidney Transplantation (Experimental): Radical nephrectomy will be used to remove a cT1a renal mass in an altruistic kidney donor. The kidney obtained from the radical nephrectomy participant with the cT1a mass removed will be transplanted to the recipient using an allograft.
  Interventions: Procedure: Donor Radical and Partial Nephrectomy; Procedure: Kidney Transplantation; Procedure: Laparoscopic Radical Nephrectomy

INTERVENTIONS:
Procedure: Donor Radical and Partial Nephrectomy — Donor participants will undergo laparoscopic radical nephrectomy (RN) . Donor kidney then will undergo cold perfusion and ex-vivo partial nephrectomy (PN) with cold ischemia. During PN, careful inspection of tumor will be performed to ensure it is well-encapsulated. If any infiltrative features (versus well encapsulated tumor) are noted intraoperatively then transplant will not be performed. Multiple surgical margins will be sent (either frozen section or standard with priority). If final margins are positive or concerning, then transplant will not be performed. Biopsies of the tumor will be performed and sent to pathology (either frozen section or standard with priority).
Procedure: Kidney Transplantation — The donor kidney will remain on ice while pathologic analysis is performed, and transplant recipient surgery is initiated (if pathologic analysis satisfactory). Cold ischemia with delay for pathology will have minimal functional impact in this setting based on extensive prior experience with renal transplantation where kidneys are routinely kept hypothermic for several hours prior to transplantation.
Procedure: Laparoscopic Radical Nephrectomy — Radical nephrectomy consists of the removal of the kidney together with the perirenal fat and regional lymph nodes. The transperitoneal approach allows early control of the renal vessels.

SUMMARY:
This study is designed to investigate a novel approach to offer more ESRD participants the benefits associated with renal transplantation by increasing the supply of available allografts

ELIGIBILITY:
Inclusion Criteria:

For Donors:

* Adults > 50 years
* Willing and able to understand and sign informed consent
* Must have high-quality pre-operative cross-sectional imaging (CT or MRI) to determine tumor characteristics and perform parenchymal volume analysis for split renal function
* Patient who is a candidate for partial nephrectomy for cT1a mass who understands that partial nephrectomy is standard of care for such mass but wishes to be an altruistic kidney donor (primary incentive is altruism) via radical nephrectomy with loss of the entire kidney.
* Functional considerations:

  o Normal baseline renal function, with eGFR > 80 ml/min/1.73 m2
  * No proteinuria on urine dipstick (negative/trace considered negative)
  * Predicted new baseline GFR (NBGFR) following radical nephrectomy would be ≥ 45
  * NBGFR would be calculated using previously described equation based on split renal function (SFR) and renal functional compensation (RFC)
  * NBGFR = global GFR x (SRFcontralateral from PVA) x 1.25 (average amount of RFC)2
* Tumor characteristics on pre-operative cross-sectional imaging:

  * Tumor appears well-encapsulated
  * Tumor appears amenable to ex-vivo partial nephrectomy with reconstruction that will leave ≥75% of the functioning parenchyma intact and well vascularized
  * Low risk of complications for the recipient after ex-vivo PN based on surgeon judgment
  * Tumor is cT1a which is defined as ≤ 4cm and confined
  * Reconstructed kidney is likely to provide NBGFR for the recipient of >30 ml/min/1.73 m2. This can be estimated as (global GFR)(SRFipsilateral) x 0.75(estimate that at least 75% of the function will be saved during ex vivo tumor excision and reconstruction). Of note most such kidneys will experience some positive functional compensation but this might be mitigated by a small amount of functional loss related to ischemia. Most studies suggest that this will really be an underestimate of the final GFR in the recipient.

For Recipients:

* Age >60
* Able to understand and willing to sign informed consent
* Presence of ESRD or CKD5 with likely progression to ESRD
* Does not have potential living donor
* Not likely to receive a more "ideal" donor kidney due to significant comorbidities and/or age

Exclusion Criteria:

For Donors:

* Known familial RCC syndrome
* Functional considerations:

  o < 50 years of age
  * Preoperative GFR < 80 ml/min/1.73 m2
  * Proteinuria on urine dipstick or urinalysis (≥1+ considered positive)
  * Predicted new baseline GFR (NBGFR) following radical nephrectomy would be < 45
  * NBGFR would be calculated using previously described equation based on split renal function (SFR) and renal functional compensation (RFC)
  * NBGFR = global GFR x (SRFcontralateral from PVA) x 1.25 (average amount of RFC)2
* Comorbidities with risk of deteriorating renal function:

  * Hypertension requiring three or more anti-hypertensives
  * Diabetes mellitus requiring insulin or with end organ damage
  * Morbid obesity
  * History of nephrolithiasis or other
* Tumor characteristics on pre-operative cross-sectional imaging:

  o Tumor has infiltrative features
  * Tumor is > 4cm (does not meet criteria for cT1a stage)
  * Regional lymphadenopathy, branch or main renal vein invasion, or other imaging findings suggestive of locally advanced disease
* Kidney characteristics on pre-operative cross-sectional imaging:

  * More than one renal artery unless can be readily and safely reconstructed
  * More than one renal vein unless can be readily and safely reconstructed
  * Duplicated collecting system unless can be readily and safely reconstructed
* High-risk features on renal mass biopsy (if obtained) or intraoperative pathology

  o Malignant non-RCC pathology

  o Rhabdoid or sarcomatoid differentiation

  o Grade 4

  o Positive or concerning margins during tumor excision
* Must be deemed appropriate living donor candidate per the standard living donor selection process at the Cleveland Clinic o All altruistic living donors undergo a complete evaluation by medical providers and social workers ensuring that they are appropriate candidates to undergo this procedure. This evaluation includes direct query into any history of psychiatric comorbidities and/or substance abuse. If present, this prompts a formal evaluation by psychiatry prior to confirmation of donor candidacy.

For Recipients:

• Traditional contraindications to kidney transplantation at the Cleveland Clinic would apply, including the following directly from the Transplant Care Pathway:

* Active, untreated bacterial, fungal, or viral infections. Once treated, patients may be reconsidered. Patients with human immunodeficiency virus (HIV)14 or chronic hepatitis15 infections will be evaluated on an individual basis.
* Active malignancy, except non-melanoma skin cancer and other selected low-grade, low-stage cancers (e.g., bladder, kidney, prostate). The American Society of Transplant (AST) clinical practice guidelines published in 2001 are dated. Improved methods of cancer prognostication are available on a cancer-specific basis.16 An acceptable disease-free waiting period may be needed prior to transplantation depending on the cancer type (stage/grade) and treatment modality. Expert opinion from an oncological specialist may be needed to facilitate decisions about wait-listing or performance of a transplant.
* Medical non-adherence, substance abuse or behaviors leading to a failure to achieve a therapeutic physician/transplant team-patient alliance.
* Life expectancy of less than five years independent of renal disease.
* Advanced circulatory disease (cardiac, cerebral, peripheral), pulmonary disease or other non-renal conditions such that transplantation would pose a significant risk for morbidity/mortality.
* Obesity with body mass index (BMI) > 38, or an abdominal wall configuration that in the judgment of the evaluating surgeon poses undue complication risk.
* Active nicotine abuse (in any form).
* Poor functional status independent of renal disease.
* Considering the average waiting times for a deceased donor kidney is more than 3 years, only transplant candidates 72 years or younger will be accepted for evaluation. Suitable candidates may remain on the waiting list up to the age of 75-year-old. They will be delisted if no transplantation has occurred.
* Cumulative burden of disease defined as multiple medical conditions that on their own may not preclude listing but that in combination are deemed not suitable by the transplant selection committee.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of Radical Nephrectomy for a Small Renal Mass | Within 30 days of surgery
  Safety and feasibility as determined by peri-operative adverse events of the following Grade 3-5 CTCAE v5.0 outcomes within 30 days of surgery:
  i. Anemia ii. Acute kidney injury
Safety and feasibility for Renal Transplant Participants Receiving a Reconstructed Donor Kidney | Within 30 days of surgery
  Safety and feasibility as determined by peri-operative adverse events of the following Grade 3-5 CTCAE v5.0 outcomes within 30 days of surgery:
  i. Anemia ii. Renal hemorrhage iii. Kidney anastomotic leak iv. Urinary fistula

SECONDARY OUTCOMES:
Surgical Outcomes for a Radical Nephrectomy for a Small Renal Mass | Within 180 days of surgery
  a. Intermediate term surgical outcomes as determined by adverse events of the following Grade 3-5 CTCAE v5.0 outcomes within 180 days of surgery: i. Anemia ii. Acute kidney injury iii. Wound infection iv. Infection and infestations - Urinary tract infection, abscess
Functional Outcomes for a Radical Nephrectomy for a Small Renal Mass | 1 year after surgery
  Renal function as determined by:
  i. Post-operative baseline GFR >45 ml/min/1.73m2 at time of follow up ii. GFR >45 ml/min/1.73m2 at one year after radical nephrectomy
Oncologic Outcomes for a Radical Nephrectomy for a Small Renal Mass | Up to 1 year after surgery
  c. Oncologic outcomes as determined by local or distant recurrence of malignancy within one year of follow up
Surgical Outcomes for a Renal Transplant Recipient After Ex-vivo Partial Nephrectomy | Within 180 days of surgery
  Intermediate term surgical outcomes as determined by adverse events of the following Grade 3-5 CTCAE v5.0 outcomes within 180 days of surgery:
  i. Anemia ii. Renal hemorrhage iii. Kidney anastomotic leak iv. Urinary fistula v. Wound infection vi. Infection and infestations - Other, Urinary tract infection, abscess, bacteremia
Functional Outcomes for a Renal Transplant Recipient After Ex-vivo Partial Nephrectomy | 1 year after surgery
  Renal function as determined by:
  i. Delayed-graft function ii. Nadir post-transplant GFR iii. GFR measured at one year follow up
Oncologic Outcomes for a Renal Transplant Recipient After Ex-vivo Partial Nephrectomy | Up to 1 year after surgery
  c. Oncologic outcomes as determined by local or distant recurrence of malignancy within one year of follow up, diagnosed by one year follow up CT imaging or other method used to determine presence of recurrent malignancy
Participant Attitudes/Decision Making Surrounding Altruistic Kidney Donation | 1 year after surgery
  Participant attitudes and decision making surrounding altruistic donation as a component of surgery for a renal mass will be determined by a survey provided to participants at a preoperative visit prior to surgery and at the 12 month follow-up visit.
Participant Attitudes/Decision Making Surrounding Transplant Recipients | 1 year after surgery
  Participant attitudes and decision-making surrounding receipt of a kidney that previously had a small renal mass will be determined by a survey provided to participants at a preoperative visit prior to surgery and at the 12-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Eltemamy, MD, Principal Investigator — Cleveland Clinic: Glickman Urological and Kidney Institute
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States